CLINICAL TRIAL: NCT03496467
Title: Clinical Study Evaluating Safety and Efficacy of a Nepafenac Punctal Plug Delivery System (N-PPDS) Compared With Placebo Punctal Plug Delivery System (p-PPDS) in Controlling Post-Operative Ocular Pain and Inflammation After Routine Unilateral Cataract Surgery
Brief Title: Safety/Efficacy of Nepafenac Punctal Plug Delivery System Compared to Placebo to Control Ocular Pain/Inflammation After Cataract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPIF-2018-01
Record Dates: First submitted 2018-03-21; First posted 2018-04-12 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Pain; Inflammation
Keywords: Treatment of pain and inflammation after Cataract Surgery
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Nepafenac PPDS (Active Comparator): N-PPDS (Nepafenac Punctal Plug Deliver System) is an L-shaped, silicone punctal plug with a drug eluting core that contains nepafenac (active)
  Interventions: Combination Product: Nepafenac PPDS
- Placebo PPDS (Placebo Comparator): p-PPDS (placebo Punctal Plug Delivery System) is an L-shaped, silicone punctal plug with a drug insert that contains no active ingredient (placebo).
  Interventions: Combination Product: Placebo PPDS

INTERVENTIONS:
Combination Product: Nepafenac PPDS — A punctal plug delivery system (PPDS) is being developed as a device that can deliver a sustained release of a drug to a specific eye. The PPDS is made up of a medical grade silicone punctal plug which holds an insert (core) that contains nepafenac, a nonsteroidal anti-inflammatory drug.
  Arms: Nepafenac PPDS
Combination Product: Placebo PPDS — A punctal plug delivery system (PPDS) is being developed as a device that can deliver a sustained release of a drug to a specific eye. The PPDS is made up of a medical grade silicone punctal plug which holds an insert (core) that does not contain nepafenac.
  Arms: Placebo PPDS

SUMMARY:
This is a Phase 2, multi-center, randomized, parallel-arm, double-masked, placebo-controlled study. One (1) to 2 days prior to their scheduled cataract surgery, each study subject will be randomized (2:1) in to one of two treatment groups: N-PPDS or p-PPDS, which are inserted in the lower punctum of the subject's scheduled surgical eye. All plugs will remain in the study subject's lower punctum for a period of 2 weeks following cataract surgery.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, parallel-arm, double-masked, placebo-controlled study. One (1) to 2 days prior to their scheduled cataract surgery, each study subject will be randomized (2:1) in to one of two treatment groups:

Group A: A total of 50 study subjects (50 eyes) will have an N-PPDS inserted in the lower punctum of their scheduled surgical eye.

Group B: A total of 25 study subjects (25 eyes) will have a p-PPDS inserted in the lower punctum of their scheduled surgical eye.

All plugs will remain in the study subject's lower punctum for a period of 2 weeks following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female subject in good general health, ≥ 22 years of age at the time of the screening visit
2. A subject with a cataract for which routine phacoemulsification extraction and implantation of an intraocular lens has been planned
3. A subject has a lower puncta that can be dilated to 1.0 mm in their scheduled surgical eye

Exclusion Criteria:

1. A subject with a history of complications, adverse events, trauma or disease in the nasolacrimal area, whether or not it was due to punctal plug wear, including but not limited to dacryocystitis, inflammation or canaliculitis in either eye
2. A subject with structural lid abnormalities (e.g., ectropion, entropion) in their schedule surgical eye
3. A subject with a puncta >0.9 mm prior to dilation in their scheduled surgical eye
4. A subject with any signs of intraocular inflammation (cells/flare) in either eye at the screening visit
5. A subject with a known sensitivity to nepafenac or any inactive ingredient of the punctum plug, silicone, fluorescein, topical anesthetic, or any other products required for study procedures or cataract surgery
6. A subject with a history of chronic/recurrent inflammatory eye disease (e.g., scleritis, uveitis, herpes keratitis) in either eye

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepank Utkhede, Study Director — Mati Therapeutics
Locations (3):
- United States (3):
  - Cincinnati Eye Institute-Edgewood, Edgewood, Kentucky
  - Ophthalmic Consultants of Long Island, Garden City, New York
  - Kerry Solomon, MD, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nepafenac PPDS | Placebo PPDS
Started | 38 | 18
Completed | 34 | 14
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac PPDS | Placebo PPDS | Total
Number analyzed (Participants) | 38 | 18 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 24 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (7.17) | 67.8 (7.64) | 67.4 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 19 | 7 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 38 | 15 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 18 | 56

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Pain
Description: Assessment of pain in subjects as measured by a scale of 0 - 5. Post-op pain scale: 0 represents absence of pain and 5 represents a definite, continuous unbearable ocular or periocular pain.
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nepafenac PPDS | Placebo PPDS
Number analyzed (Participants) | 34 | 14
Participants
  no pain | 30 | 13
  trace pain | 2 | 0
  mild pain | 2 | 1
  moderate pain | 0 | 0
  severe pain | 0 | 0
  intolerable pain | 0 | 0

2. Secondary Outcome: Assessment of Anterior Chamber Cells
Description: Anterior chamber cells are assessed using a scale of 0 - 4 with 0 representing no cells seen and 4 representing >30 cells seen.
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nepafenac PPDS | Placebo PPDS
Number analyzed (Participants) | 34 | 14
Participants
  None: no cells seen | 22 | 7
  Trace: 1-5 cells seen | 7 | 3
  Mild: 6-15 cells seen | 5 | 4
  Moderate: 16-30 cells seen | 0 | 0
  Severe: >30 cells seen | 0 | 0

3. Secondary Outcome: Assessment of Flare
Description: Anterior chamber flare is assessed using a scale of 0 - 4 with 0 representing no Tyndall effect and 4 representing Tyndall effect in anterior chamber is very intense
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nepafenac PPDS | Placebo PPDS
Number analyzed (Participants) | 34 | 14
Participants
  None: No Tyndall effect | 29 | 10
  Trace: Tyndall effect barely discernible | 3 | 1
  Mild: Tyndall effect in anterior chamber is clearly visible | 2 | 3
  Moderate: Tyndall effect in anterior chamber is moderately intense | 0 | 0
  Severe: Tyndall effect in anterior chamber is very intense. The aqueous has a white milky appearance | 0 | 0

ADVERSE EVENTS:
Time Frame: The Nepafenac PPDS or Placebo PPDS was inserted 1-2 days prior to surgery. Subjects were followed for 14 days (+/-2 days) post op
Description: Subjects were asked: "Have you had any problems since your last visit?"
Arm/Group | Nepafenac PPDS | Placebo PPDS
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/18
Other Adverse Events (participants affected / at risk) | 10/38 | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nepafenac PPDS (N=38) | Placebo PPDS (N=18)
elevated IOP (Eye disorders) | 3 (3) | 0 (0)
iritis (Eye disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
posterior capsule rupture (Eye disorders) | 0 (0) | 1 (1)
Cavity, 3rd molar (General disorders) | 1 (1) | 0 (0)
Pain/irritation/inflammation (Eye disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT03496467/Prot_SAP_000.pdf